CLINICAL TRIAL: NCT04382066
Title: Multicenter, Randomized, Parallel and Proof of Concept Study to Evaluate the Safety Profile of Three Doses of Plitidepsin in Patients With COVID-19 Requiring Hospitalization
Brief Title: Proof of Concept Study to Evaluate the Safety Profile of Plitidepsin in Patients With COVID-19
Acronym: APLICOV-PC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL-D-002-20; 2020-001993-31 (EudraCT Number)
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Plitidepsin; COVID-19; SARS-COV-2; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): Plitidepsin 1.5 mg / day x 3 consecutive days
  Interventions: Drug: Plitidepsin 1.5 mg/day
- Experimental 2 (Experimental): Plitidepsin 2.0 mg / day x 3 consecutive days
  Interventions: Drug: Plitidepsin 2.0 mg/day
- Experimental 3 (Experimental): Plitidepsin 2.5 mg / day x 3 consecutive days
  Interventions: Drug: Plitidepsin 2.5 mg/day

INTERVENTIONS:
Drug: Plitidepsin 1.5 mg/day — Plitidepsin 1.5 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
  All patients must receive the following prophylactic medications 20-30 minutes before the infusion of plitidepsin:
  * Diphenhydramine hydrochloride 25 mg iv or equivalent.
  * Ranitidine 50 mg iv or equivalent.
  * Dexamethasone 8 mg iv.
  * Ondansetron 8 mg i.v. 15 minutes infusion or equivalent.
  * Ondansetron 4 mg p.o. administered every 12 hours until 48 hours after the last administration of plitidepsin.
  Arms: Experimental 1
Drug: Plitidepsin 2.0 mg/day — Plitidepsin 2.0 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
  All patients must receive the following prophylactic medications 20-30 minutes before the infusion of plitidepsin:
  * Diphenhydramine hydrochloride 25 mg iv or equivalent.
  * Ranitidine 50 mg iv or equivalent.
  * Dexamethasone 8 mg iv.
  * Ondansetron 8 mg i.v. 15 minutes infusion or equivalent.
  * Ondansetron 4 mg p.o. administered every 12 hours until 48 hours after the last administration of plitidepsin.
  Arms: Experimental 2
Drug: Plitidepsin 2.5 mg/day — Plitidepsin 2.5 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
  All patients must receive the following prophylactic medications 20-30 minutes before the infusion of plitidepsin:
  * Diphenhydramine hydrochloride 25 mg iv or equivalent.
  * Ranitidine 50 mg iv or equivalent.
  * Dexamethasone 8 mg iv.
  * Ondansetron 8 mg i.v. 15 minutes infusion or equivalent.
  * Ondansetron 4 mg p.o. administered every 12 hours until 48 hours after the last administration of plitidepsin.
  Arms: Experimental 3

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (SARS-CoV-2) from these pneumonia patients and developed a real-time reverse transcription PCR (real-time RT-PCR) diagnostic assay.

Given no specific antiviral therapy for COVID-19 and the ready availability of plitidepsin as a potential antiviral agent, based on pre-clinical studies, this randomized, parallel and proof of concept trial will evaluate the safety of three doses of plitidepsin in patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
In December 2019, a new infectious respiratory disease emerged in Wuhan, China. The agent that caused this pneumonia was identified as a new virus in the Coronaviridae family (SARS-CoV-2) and the clinical symptomatology associated with the virus has been named COVID-19. COVID-19 is currently a public health emergency.

Plitidepsin is an authorized drug in Australia for the treatment of multiple myeloma. Antiviral activity of plitidepsin has been analyzed in a human hepatoma cell line infected with the HCoV-229E-GFP virus, a virus similar to the SARS-CoV-2 virus.

Taking into account that the available safety data from plitidepsin comes from patients with solid tumors that received treatment with a regimen of administration of plitidepsin for 5 consecutive days, we propose a multicenter, randomized, proof-of-concept clinical trial to assess the safety profile of 3 different dose levels of plitidepsin administered three consecutive days, in adult patients with confirmed diagnosis of COVID-19 who require hospital admission.

This study aims to assess safety and toxicity profile and also preliminary efficacy of plitidepsin at each dose level administered according to the proposed administration scheme in patients with COVID-19 who require hospital admission. Main objective is to select the recommended dose levels of plitidepsin for a future phase II / III efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who agrees to participate in the study by signing the informed consent.
2. Men and women (non-pregnant) aged ≥18 years.
3. COVID-19 infection confirmed by PCR obtained from nasopharyngeal exudate or sample from the lower respiratory tract.
4. Patients who require hospitalization for COVID-19.
5. Symptom onset at most within 10 days prior to study inclusion.
6. Men and women with reproductive capacity should agree to use highly effective contraceptive methods during their participation in the study and in the 6 months following the last administration of plitidepsin.
7. In addition, women participating in the study with reproductive ability must have a negative pregnancy test at enrollment.

Exclusion Criteria:

1. Patients participating in some other clinical trial for COVID-19 infection.
2. Patients who are receiving treatment with antivirals, interleukin 6 receptor inhibitors or immunomodulatory drugs for COVID-19.
3. Patients who are receiving treatment with chloroquine and derivatives.
4. Evidence of multi-organ failure.
5. Patients who require support with mechanical ventilation (invasive or non-invasive) at the time of inclusion.
6. D-dimer> 4 x UNL.
7. Hb <9 g / dL.
8. Neutrophils <1000 / mm3.
9. Platelets <100,000 / mm3.
10. Lymphopenia <800 / μL.
11. GOT / GPT> 3 X UNL.
12. Bilirubin> 1 X UNL.
13. CPK> 2.5 X UNL.
14. Creatinine clearance <30ml / min.
15. Troponin elevation> 1.5 x ULN.
16. Clinically relevant heart disease (NYHA> 2).
17. Clinically relevant arrhythmia or previous history / presence of prolonged QT-QTc ≥ 450 ms.
18. Pre-existing neuropathies of any type ≥ grade 2.
19. Hypersensitivity to the active substance or to any of its excipients (macrogol glycerol ricinoleate and ethanol).
20. Patients who require or are being treated with potent CYP3A4 inhibitors and inducers.
21. Patients who for any reason should not be included in the study according to the evaluation of the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Estrada, MD, Principal Investigator — Hospital San Carlos, Madrid; Jesús Fortún, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; José Barberán, MD, Principal Investigator — HOSPITAL UNIVERSITARIO HM MONTEPRÍNCIPE
Locations (13):
- Spain (13):
  - Hospital Universitario Hm Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Ciudad Real, Ciudad Real
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital La Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hosptial Quironsalud Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Data of the final publication of the study will be shared upon request.

REFERENCES:
- [Derived] Varona JF, Landete P, Lopez-Martin JA, Estrada V, Paredes R, Guisado-Vasco P, Fernandez de Orueta L, Torralba M, Fortun J, Vates R, Barberan J, Clotet B, Ancochea J, Carnevali D, Cabello N, Porras L, Gijon P, Monereo A, Abad D, Zuniga S, Sola I, Rodon J, Vergara-Alert J, Izquierdo-Useros N, Fudio S, Pontes MJ, de Rivas B, Giron de Velasco P, Nieto A, Gomez J, Aviles P, Lubomirov R, Belgrano A, Sopesen B, White KM, Rosales R, Yildiz S, Reuschl AK, Thorne LG, Jolly C, Towers GJ, Zuliani-Alvarez L, Bouhaddou M, Obernier K, McGovern BL, Rodriguez ML, Enjuanes L, Fernandez-Sousa JM, Krogan NJ, Jimeno JM, Garcia-Sastre A. Preclinical and randomized phase I studies of plitidepsin in adults hospitalized with COVID-19. Life Sci Alliance. 2022 Jan 10;5(4):e202101200. doi: 10.26508/lsa.202101200. Print 2022 Apr. PMID 35012962

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental 1: Plitidepsin 1.5 mg / day x 3 consecutive days
  Plitidepsin 1.5 mg/day: Plitidepsin 1.5 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
- Experimental 2: Plitidepsin 2.0 mg / day x 3 consecutive days
  Plitidepsin 2.0 mg/day: Plitidepsin 2.0 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
- Experimental 3: Plitidepsin 2.5 mg / day x 3 consecutive days
  Plitidepsin 2.5 mg/day: Plitidepsin 2.5 mg/day will be IV infused through a pump device over 1 hour and 30 minutes, 3 consecutive days.
Period: Overall Study
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3
Started (One patient withdrew the Informed Consent before any study procedure was performed.) | 15 | 15 | 15
Completed 3-day Treatment | 14 | 15 | 15
Completed (Completed Day 31 follow-up) | 13 | 15 | 14
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 11 | 36
  >=65 years | 3 | 2 | 4 | 9
Age, Continuous [Median (Full Range); unit: years] | 51 [32 to 75] | 49 [34 to 71] | 53 [31 to 84] | 52 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 15
  Male | 11 | 11 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 15 | 15 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 15 | 45
Number of comorbidities [Number; unit: Participants]
  None | 5 | 2 | 2 | 9
  One | 2 | 7 | 6 | 15
  Two or more | 8 | 6 | 7 | 21
Comorbidities [Number; unit: Participants]
  Cardiac disease | 1 | 0 | 1 | 2
  Kidney disease | 0 | 1 | 0 | 1
  Lung disease (COPD) | 1 | 1 | 1 | 3
  Asthma | 2 | 0 | 3 | 5
  Diabetes | 1 | 5 | 2 | 8
  Hypertension | 2 | 2 | 5 | 9
  Obesity | 1 | 5 | 4 | 10
Clinical status at randomization [Number; unit: Participants]
  Mild COVID-19 infection | 2 | 3 | 1 | 6
  Moderate COVID-19 infection | 8 | 7 | 8 | 23
  Severe COVID-19 infection | 5 | 5 | 6 | 16
Chest x-rays [Number; unit: Participants]
  Abnormal | 15 | 13 | 13 | 41
  Bilateral pneumonia | 11 | 10 | 11 | 32
Body temperature [Median (Full Range); unit: Degrees Celsius] | 36.5 [35.0 to 39.1] | 37.0 [35.0 to 38.9] | 36.2 [35.0 to 38.0] | 36.5 [35.0 to 39.1]
Systolic blood pressure [Median (Full Range); unit: mmHg] | 113 [99 to 132] | 115 [90 to 130] | 124 [98 to 150] | 119 [90 to 150]
Diastolic blood pressure [Median (Full Range); unit: mmHg] | 69 [59 to 85] | 71 [50 to 90] | 78 [57 to 88] | 72 [50 to 90]
Heart rate [Median (Full Range); unit: Bpm] | 84 [62 to 107] | 78 [60 to 120] | 82 [57 to 100] | 82 [57 to 120]
Respiratory rate [Median (Full Range); unit: Bpm] | 17 [14 to 24] | 18 [14 to 24] | 16.5 [12 to 26] | 17 [12 to 26]
Oxygen saturation at room air [Median (Full Range); unit: Percentage] — Population: Oxygen saturation at room air has been analyzed for the 22 patients who did not requiere supplementary O2.
  Percentage
    number analyzed (Participants) | 9 | 7 | 6 | 22
    (all) | 95 [92 to 99] | 95 [91 to 97] | 96.5 [94 to 97] | 95.5 [91 to 99]
On supplementary O2 [Number; unit: Participants] | 6 | 8 | 9 | 23
PaO2/FiO2 [Median (Full Range); unit: Ratio] | 358 [336 to 408] | 352 [285 to 396] | 343 [253 to 481] | 350 [253 to 481]
White Blood Cells (WBC) [Median (Full Range); unit: 10^9 cells/liter] | 4.4 [2.6 to 7.3] | 5.4 [3.3 to 8.4] | 7.1 [4.0 to 16.0] | 5.5 [2.6 to 16.0]
Platelet count [Median (Full Range); unit: 10^9 cells/liter] | 183 [118 to 362] | 168 [127 to 339] | 244 [108 to 462] | 183 [108 to 462]
Lymphocytes [Median (Full Range); unit: 10^9 cells/liter] | 0.9 [0.8 to 2.1] | 1.1 [0.6 to 1.5] | 1.1 [0.7 to 3.0] | 1.0 [0.6 to 3.0]
D-dimer [Median (Full Range); unit: ng/mL] | 330 [162 to 1081] | 463 [200 to 1270] | 415 [106 to 962] | 405 [106 to 1270]
Ferritin [Median (Full Range); unit: ng/ml] | 408 [96.8 to 1652.8] | 597 [174 to 1055.2] | 363 [12.2 to 1647] | 412 [12.2 to 1652.8]
C-reactive protein [Median (Full Range); unit: mg/L] | 17.7 [1.2 to 120.4] | 67.2 [2.1 to 128.0] | 32.6 [0.3 to 120.0] | 32.7 [0.3 to 128.0]
Serum creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.8 [0.6 to 1.4] | 0.8 [0.5 to 1.2] | 0.8 [0.6 to 1.2] | 0.8 [0.5 to 1.4]
Alanine aminotransferase [Median (Full Range); unit: x Upper Limit of Normal (ULN)] | 0.9 [0.3 to 1.9] | 0.8 [0.4 to 1.7] | 0.7 [0.2 to 1.8] | 0.8 [0.2 to 1.9]
Aspartate aminotransferase [Median (Full Range); unit: x Upper Limit of Normal (ULN)] | 0.8 [0.4 to 1.5] | 0.9 [0.5 to 1.7] | 0.7 [0.3 to 2.4] | 0.8 [0.3 to 2.4]
Lactate dehydrogenase [Median (Full Range); unit: x Upper Limit of Normal (ULN)] | 1.0 [0.7 to 1.7] | 1.0 [0.8 to 2.0] | 1.2 [0.5 to 1.4] | 1.0 [0.5 to 2.0]
Creatine phosphokinase [Median (Full Range); unit: x Upper Limit of Normal (ULN)] | 0.4 [0.1 to 2.7] | 0.3 [0.2 to 1.7] | 0.4 [0.1 to 4.0] | 0.4 [0.1 to 4.0]
Viral load [Median (Full Range); unit: Log10 copies/mL] — Population: Results available por 44 patients: 1 patient (in 2.0 mg cohort) did not have baseline viral load asessment by central lab.
  Log10 copies/mL
    number analyzed (Participants) | 15 | 14 | 15 | 44
    (all) | 6.3 [1.5 to 9.7] | 6.2 [3.8 to 7.0] | 5.7 [1.5 to 10.6] | 6.1 [1.5 to 10.6]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Occurrence of Neutropenia ≥ Grade 3
Description: Percentage of patients with Neutropenia ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Groups:
- Total: All the 45 patients treated with at least 1 dose of plitidepsin were analyzed for safety.
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

2. Primary Outcome: Frequency of Occurrence of Thrombocytopenia ≥ Grade 3
Description: Percentage of patients with Thrombocytopenia ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

3. Primary Outcome: Frequency of Occurrence of Anemia ≥ Grade 3
Description: Percentage of patients with Anemia ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

4. Primary Outcome: Frequency of Occurrence of Lymphopenia ≥ Grade 3
Description: Percentage of patients with Lymphopenia ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

5. Primary Outcome: Frequency of Occurrence of CPK Increase ≥ Grade 3
Description: Percentage of patients with CPK increase ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

6. Primary Outcome: Frequency of Occurrence of Increase ALT and / or AST ≥ Grade 3
Description: Percentage of patients with Increase ALT and / or AST ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  ALT increased Day 3 | 0 | 0 | 0 | 0
  ALT increased Day 7 | 0 | 0 | 0 | 0
  ALT increased Day 15 | 0 | 1 | 0 | 1
  ALT increased Day 31 | 0 | 1 | 0 | 1
  AST increased Day 3 | 0 | 0 | 0 | 0
  AST increased Day 7 | 0 | 0 | 0 | 0
  AST increased Day 15 | 0 | 0 | 0 | 0
  AST increased Day 31 | 0 | 0 | 0 | 0

7. Primary Outcome: Frequency of Occurrence of Increase Total Bilirubin or Direct Bilirubin ≥ Grade 3
Description: Percentage of patients with Increase total bilirubin or direct bilirubin ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

8. Primary Outcome: Frequency of Occurrence of Neurotoxicity ≥ Grade 3
Description: Percentage of patients with Neurotoxicity ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

9. Primary Outcome: Frequency of Occurrence of QT-QTc Interval Extension ≥ Grade 3
Description: Percentage of patients with QT-QTc interval extension ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 0 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 0 | 0 | 0 | 0

10. Primary Outcome: Frequency of Occurrence of Other Adverse Events ≥ Grade 3
Description: Percentage of patients with Other adverse events ≥ grade 3 according to NCI-CTCAE v5.0 criteria.
Time Frame: At days 3, 7, 15 and 31.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Leukocytosis day 3 | 0 | 0 | 1 | 1
  Leukocytosis day 7 | 0 | 0 | 1 | 1
  Leukocytosis day 15 | 0 | 0 | 1 | 1
  Leukocytosis day 31 | 0 | 0 | 1 | 1
  Diarrhoea day 3 | 0 | 0 | 1 | 1
  Diarrhoea day 7 | 0 | 0 | 1 | 1
  Diarrhoea day 15 | 0 | 0 | 1 | 1
  Diarrhoea day 31 | 0 | 0 | 1 | 1
  Condition aggravated day 3 | 1 | 0 | 0 | 1
  Condition aggravated day 7 | 1 | 0 | 0 | 1
  Condition aggravated day 15 | 1 | 0 | 0 | 1
  Condition aggravated day 31 | 1 | 0 | 0 | 1
  Anaphylactic reaction day 3 | 1 | 0 | 0 | 1
  Anaphylactic reaction day 7 | 1 | 0 | 0 | 1
  Anaphylactic reaction day 15 | 1 | 0 | 0 | 1
  Anaphylactic reaction day 31 | 1 | 0 | 0 | 1
  Bacteraemia day 3 | 0 | 0 | 0 | 0
  Bacteraemia day 7 | 0 | 0 | 1 | 1
  Bacteraemia day 15 | 0 | 0 | 1 | 1
  Bacteraemia day 31 | 0 | 0 | 1 | 1
  COVID-19 pneumonia day 3 | 0 | 0 | 0 | 0
  COVID-19 pneumonia day 7 | 0 | 0 | 1 | 1
  COVID-19 pneumonia day 15 | 1 | 0 | 1 | 2
  COVID-19 pneumonia day 31 | 1 | 0 | 1 | 2
  Pneumonia day 3 | 0 | 0 | 0 | 0
  Pneumonia day 7 | 0 | 0 | 0 | 0
  Pneumonia day 15 | 1 | 0 | 0 | 1
  Pneumonia day 31 | 1 | 0 | 0 | 1
  Superinfection bacterial day 3 | 0 | 0 | 0 | 0
  Superinfection bacterial day 7 | 0 | 0 | 0 | 0
  Superinfection bacterial day 15 | 0 | 0 | 0 | 0
  Superinfection bacterial day 31 | 0 | 0 | 1 | 1
  Urinary tract infection day 3 | 0 | 0 | 0 | 0
  Urinary tract infection day 7 | 0 | 0 | 1 | 1
  Urinary tract infection day 15 | 0 | 0 | 1 | 1
  Urinary tract infection day 31 | 0 | 0 | 1 | 1
  C-reactive protein increased day 3 | 0 | 0 | 0 | 0
  C-reactive protein increased day 7 | 1 | 0 | 0 | 1
  C-reactive protein increased day 15 | 1 | 0 | 0 | 1
  C-reactive protein increased day 31 | 1 | 0 | 0 | 1
  Gamma-glutamyltransferase increased day 3 | 0 | 1 | 0 | 1
  Gamma-glutamyltransferase increased day 7 | 1 | 1 | 0 | 2
  Gamma-glutamyltransferase increased day 15 | 1 | 2 | 0 | 3
  Gamma-glutamyltransferase increased day 31 | 1 | 2 | 0 | 3
  Serum ferritin increased day 3 | 0 | 0 | 0 | 0
  Serum ferritin increased day 7 | 1 | 0 | 0 | 1
  Serum ferritin increased day 15 | 1 | 0 | 0 | 1
  Serum ferritin increased day 31 | 1 | 0 | 0 | 1
  Hyperglycaemia day 3 | 0 | 0 | 1 | 1
  Hyperglycaemia day 7 | 0 | 0 | 1 | 1
  Hyperglycaemia day 15 | 0 | 0 | 1 | 1
  Hyperglycaemia day 31 | 0 | 0 | 1 | 1
  Status epilepticus day 3 | 0 | 0 | 0 | 0
  Status epilepticus day 7 | 0 | 0 | 0 | 0
  Status epilepticus day 15 | 0 | 0 | 0 | 0
  Status epilepticus day 31 | 0 | 0 | 1 | 1
  Acute respiratory distress syndrome day 3 | 0 | 0 | 0 | 0
  Acute respiratory distress syndrome day 7 | 1 | 1 | 0 | 2
  Acute respiratory distress syndrome day 15 | 1 | 1 | 1 | 3
  Acute respiratory distress syndrome day 31 | 2 | 1 | 1 | 4
  Pneumomediastinum day 3 | 0 | 0 | 0 | 0
  Pneumomediastinum day 7 | 0 | 0 | 0 | 0
  Pneumomediastinum day 15 | 0 | 0 | 0 | 0
  Pneumomediastinum day 31 | 0 | 0 | 1 | 1
  Respiratory distress day 3 | 0 | 0 | 0 | 0
  Respiratory distress day 7 | 0 | 0 | 1 | 1
  Respiratory distress day 15 | 0 | 0 | 1 | 1
  Respiratory distress day 31 | 0 | 0 | 1 | 1

11. Primary Outcome: Percentage of Patients in Whom Treatment Cannot be Completed.
Description: Percentage of patients in whom treatment cannot be completed and the reasons.
Time Frame: At 3 days from the first dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants | 1 | 0 | 0 | 1

12. Primary Outcome: Percentage of Patients With Adverse Events.
Description: Percentage of patients with adverse events.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 14 | 11 | 13 | 38
  Day 7 | 15 | 14 | 15 | 44
  Day 15 | 15 | 14 | 15 | 44
  Day 31 | 15 | 14 | 15 | 44

13. Primary Outcome: Percentage of Patients With Serious Adverse Events.
Description: Percentage of patients with serious adverse events.
Time Frame: At days 3, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 3 | 1 | 0 | 0 | 1
  Day 7 | 4 | 1 | 0 | 5
  Day 15 | 4 | 1 | 2 | 7
  Day 31 | 6 | 1 | 3 | 10

14. Primary Outcome: Percentage of Patients With ECG Abnormalities.
Description: Percentage of patients with ECG abnormalities.
Time Frame: At days 2, 3, 4, 5, 6, 7, 15 and 31
Measure: Count of Participants; unit: Participants
Groups:
- Experimental 1: Plitidepsin 1.5 mg & day x 3 consecutive days
- Experimental 2: Plitidepsin 2.0 mg & day x 3 consecutive days
- Experimental 3: Plitidepsin 2.5 mg & day x 3 consecutive days
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Participants
  Day 2 | 2 | 3 | 3 | 8
  Day 3 | 4 | 2 | 2 | 8
  Day 4 | 3 | 1 | 1 | 5
  Day 5 | 3 | 1 | 2 | 6
  Day 6 | 4 | 1 | 2 | 7
  Day 7 | 1 | 1 | 3 | 5
  Day 15 | 2 | 2 | 2 | 6
  Day 31 | 2 | 0 | 1 | 3

15. Secondary Outcome: Change in the Viral Load of SARS-CoV-2
Description: Median change in the viral load of SARS-CoV-2 from baseline.
Time Frame: At days 4, 7, 15 and 31
Population: One patient dosed at 1.5 mg experienced an anaphylactic reaction during the first plitidepsin infusion and discontinued study treatment, so was not considered evaluable for efficacy.
Measure: Median (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Log10 copies/mL
  Day 4 | -1.23 (1.30) | -1.49 (1.42) | -1.32 (1.90) | -1.35 (1.54)
  Day 7 | -2.55 (1.65) | -2.26 (1.68) | -2.25 (1.61) | -2.35 (1.61)
  Day 15 | -4.22 (2.58) | -2.70 (2.23) | -2.92 (1.91) | -3.25 (2.29)
  Day 31 | -4.70 (1.74) | -3.53 (2.07) | -3.49 (2.94) | -3.85 (2.35)

16. Secondary Outcome: Time to Negative PCR Test for COVID-19
Description: Time from inclusion/randomization to date of negative PCR test for COVID-19
Time Frame: Up to 31 days + 3 days for window period
Population: as for outcome 15
Measure: Mean (Full Range); unit: Days
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Days | 11 [3 to 29] | 14 [3 to 30] | 14 [3 to 33] | 13 [3 to 33]

17. Secondary Outcome: Mortality
Description: Percentage of patients who die during the study
Time Frame: At days 7, 15 and 31
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Participants
  Day 7 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0
  Day 31 | 1 | 0 | 1 | 2

18. Secondary Outcome: Percentage of Patients Requiring Invasive Mechanical Ventilation and / or ICU Admission
Description: Percentage of patients requiring invasive mechanical ventilation and / or ICU admission
Time Frame: At days 7, 15 and 31
Population: One patient dosed at 1.5 mg experienced an anaphylactic reaction during the first plitidepsin infusion and discontinued study treatment, so was not considered evaluable for efficacy. Cumulative results.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Participants
  Day 7 | 2 | 1 | 2 | 5
  Day 15 | 2 | 1 | 3 | 6
  Day 31 | 2 | 1 | 3 | 6

19. Secondary Outcome: Percentage of Patients Requiring Non-invasive Mechanical Ventilation
Description: Percentage of patients requiring non-invasive mechanical ventilation
Time Frame: At days 7, 15 and 31
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Participants
  Day 7 | 4 | 0 | 1 | 5
  Day 15 | 5 | 0 | 2 | 7
  Day 31 | 5 | 1 | 2 | 8

20. Secondary Outcome: Percentage of Patients Requiring Oxygen Therapy
Description: Percentage of patients requiring oxygen therapy
Time Frame: At days 7, 15 and 31
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
Number analyzed (Participants) | 14 | 15 | 15 | 44
Participants
  Day 7 | 12 | 12 | 11 | 35
  Day 15 | 12 | 12 | 11 | 35
  Day 31 | 12 | 12 | 11 | 35

ADVERSE EVENTS:
Time Frame: From first administration of plitidepsin until day 31.
Description: 2 patients die during the study, one of Arm A on day 22 due to COVID-19 pneumonia and pneumomediastinum and the other of Arm C at day 30 due to disease-related acute respiratory distress syndrome.
Arm/Group | Experimental 1 | Experimental 2 | Experimental 3 | Total
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/15 | 1/15 | 2/45
Serious Adverse Events (participants affected / at risk) | 6/15 | 1/15 | 3/15 | 10/45
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15 | 15/15 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental 1 (N=15) | Experimental 2 (N=15) | Experimental 3 (N=15) | Total (N=45)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Anaphylactic reaction Grade 3 in Arm A (1.5 mg plitidepsin) attributed to plitidepsin.
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1) | 4 (5) — 1 Acute respiratory distress syndrome grade 3 and 1 grade 4 and 1 grade 5 in the same patient in Arm A (1.5 mg plitidepsin), 1 grade 4 in Arm B (2 mg plitidepsin) and 1 grade 4 in Arm C (2.5 mg plitidepsin).
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) — Acute respiratory failure grade 5 in Arm C (2.5 mg plitidepsin)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Status epilepticus grade 3 in Arm C (2.5 mg plitidepsin)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Condition aggravated grade 3 in Arm A (1.5 mg plitidepsin)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 2 (3) — 1 COVID-19 pneumonia grade 3 in Arm A (1.5 mg ) and 1 grade 3 and 1 grade 5 in the same patient in Arm C (2.5 mg plitidepsin).
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental 1 (N=15) | Experimental 2 (N=15) | Experimental 3 (N=15) | Total (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) — 1 Leukocytosis grade 3 in Arm C (2.5 mg plitidepsin).
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 1 (1) | 3 (5)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (6) | 3 (3) | 8 (10) — 1 diarrhoea grade 3 in Arm A (1.5 mg plitidepsin) was attributed to plitidepsin.
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (9) | 6 (7) | 7 (9) | 19 (25)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (7) | 8 (12)
Hypoalbuminaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — 1 Bacteremia grade 3 in Arm C (2.5 mg plitidepsin).
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) — 1 Pneumonia grade 3 in Arm A (1.5 mg plitidepsin).
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — 1 Urinary tract infection grade 3 in Arm C (2.5 mg plitidepsin).
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
ALT increased (Investigations) | 2 (4) | 1 (3) | 2 (2) | 5 (9) — 1 ALT increased grade 3 in Arm B (2 mg plitidepsin).
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
AST increased (Investigations) | 1 (2) | 1 (2) | 1 (1) | 3 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 4 (8) | 4 (4) | 3 (4) | 11 (16) — 1 C-reactive protein increased grade 3 in Arm A (1.5 mg plitidepsin).
Ferritin increased (Investigations) | 5 (11) | 4 (6) | 5 (5) | 14 (22) — 1 Ferritin increased grade 3 in Arm A (1.5 mg plitidepsin).
GGT increased (Investigations) | 3 (8) | 2 (5) | 1 (1) | 6 (14) — 1 GGT increased grade 3 in Arm A (1.5 mg plitidepsin) and 2 grade 3 in Arm B (2 mg plitidepsin)
LDH increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
LDL increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Triglycerides increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fibrin D dimer increased (Investigations) | 3 (5) | 2 (3) | 3 (3) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 3 (7) | 8 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 0 (0) | 6 (8)
Insomnia (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 4 (5)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) — 1 Renal impairment grade 3 in Arm A (1.5 mg plitidepsin).
Breast engorgement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 4 (5) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Phlebitis (Vascular disorders) | 3 (3) | 3 (5) | 2 (2) | 8 (10)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (4) | 1 (3) | 2 (3) | 6 (10)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (10) | 5 (12) | 7 (17) | 20 (39)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Interleukin level increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of patients. No control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT04382066/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04382066/SAP_001.pdf